CLINICAL TRIAL: NCT03965637
Title: Effect of Ascorbic Acid Administration on Intraoperative Blood Loss and Wound Healing in Total Abdominal Hysterectomy
Brief Title: Intravenous Ascorbic Acid Administration in Hysterectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Zahra Vahdat Shariatpanahi, Associate Professor, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17912
Record Dates: First submitted 2019-05-26; First posted 2019-05-29 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Abdominal Hysterectomy
Keywords: vitamin c; Hysterectomy; bleeding; wound healing; abdominal surgeries
MeSH Terms: conditions — Hemorrhage | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vitamin C (Experimental): Intervention patients will be received double dose of Ascorbic acid via intravenous injection
  Interventions: Drug: vitamin C
- Control (No Intervention): Control patients will not be received any intervention

INTERVENTIONS:
Drug: vitamin C — water-soluble vitamin C injection contain of 1000 mg vitamin C that given via intravenous injection
  Other Names: ascorbic acid
  Arms: vitamin C

SUMMARY:
vitamin C or ascorbic acid has known role in tissue repair. due to it's properties(water_soluble), vitamin c is not stored in the body and when depleted, the bleeding tendency will increase due to dysfunctional connective tissues production in vessel wall and it has some important functions in platelets.

DETAILED DESCRIPTION:
In this randomized clinical trial, 1000 mg vitamin C will administrate intravenously a day before surgery and during surgery in patients who undergo abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* To be 18 years and older
* No smoking
* No history of bleeding disorder
* No history of favism
* No history of uterus, ovary, cervical cancer

Exclusion Criteria:

* Need to injection of vasopressor drugs
* Surgeon disagreement

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
volume of hemorrhage | During surgery
  volume of hemorrhage during surgery

SECONDARY OUTCOMES:
Hemoglobin value | 6 and 24 hours after surgery
  Hemoglobin value after surgery
wound healing | during 2 weeks post surgery
  complications after surgery
duration of stay in hospital | up to 2 weeks post surgery
  Length of stay in hospital
Infection | up to 2 weeks post surgery
  Developing infection up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: zahra vahdat shariatpanahi, MD,PhD, Study Chair — Associatec professor
Locations (1):
- Faculty of Nutrition and Food Technology, Shahid Beheshti University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farahani-Jam S, Yaghmaei M, Vahdat Shariatpanahi Z. Effect of intravenous ascorbic acid administration on hemorrhage and wound complications in total abdominal hysterectomy: A prospective randomized clinical trial. Clin Nutr ESPEN. 2022 Jun;49:74-78. doi: 10.1016/j.clnesp.2022.03.024. Epub 2022 Mar 26. PMID 35623878